CLINICAL TRIAL: NCT07407816
Title: Feasibility Study of the Supira System in Patients Undergoing High-Risk Percutaneous Coronary Intervention (HRPCI) Who May Benefit From Mechanical Circulatory Support Beyond the PCI Procedure
Brief Title: Study of the Supira System in Patients With Complex High-Risk Percutaneous Coronary Intervention (HRPCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Supira Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-10005
Record Dates: First submitted 2026-01-31; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Disease; Coronary Arterial Disease (CAD); Heart Failure
Keywords: Percutanous ventricular assist device; Supira System
MeSH Terms: conditions — Heart Diseases; Heart Failure

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRPCI with low LVEF and severe CAD (Experimental): Patients undergoing HRPCI with low LVEF and severe coronary artery disease who may benefit from cardiovascular hemodynamic support beyond the PCI procedure
  Interventions: Device: Supira System

INTERVENTIONS:
Device: Supira System — The Supira System is a minimally invasive, percutaneous ventricular assist device (pVAD) that is intended to provide hemodynamic support to patients undergoing high risk percutaneous coronary intervention (HRPCI). The Catheter is inserted percutaneously via the femoral artery, across the aortic valve, and into the left ventricle under fluoroscopic guidance. The left ventricle is unloaded by pumping blood from the ventricle into the ascending aorta and systemic circulation.

SUMMARY:
The objective of this study is to assess the safety and feasibility of the Supira System in heart failure patients with low LVEF, undergoing HRPCI with use of mechanical circulatory support who may benefit from cardiovascular hemodynamic support beyond the PCI procedure.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, single-arm, multi-center, feasibility study.

The Supira System is a minimally invasive, percutaneous ventricular assist device (pVAD) that is intended to provide hemodynamic support to patients undergoing high risk percutaneous coronary intervention (HRPCI) and requiring hemodynamic support. The Catheter is inserted percutaneously, across the aortic valve, and into the left ventricle under fluoroscopic guidance. The left ventricle is unloaded by pumping blood from the ventricle into the ascending aorta and systemic circulation.

ELIGIBILITY:
Inclusion Criteria:

* Subject has pre-existing heart failure, with NYHA Class II, III or IV prior to the index admission and documented LVEF ≤ 45%
* Subject is presenting with one of the following criteria: unprotected left main coronary artery (ULMCA) disease, last patent vessel, or 3-vessel disease
* Subject may benefit from hemodynamic support beyond the index procedure
* Informed consent granted by the patient or legally authorized representative

Exclusion Criteria:

* Stroke within 6 months of the index procedure, or any prior stroke with permanent neurologic deficit
* Aortic valvular disease or regurgitation categorized as moderate or greater (≥2+ on a 4-grade scale as assessed on TTE)
* Aortic stenosis and/or aortic regurgitation categorized as moderate or greater (mean gradient >20 mmHg or valve area <1.5 cm2 as assessed on TTE)
* Presence of decompensated liver disease; severe liver dysfunction (Child-Pugh Score class C)
* Ongoing renal replacement therapy with dialysis or continues renal replacement therapy
* Heparin-induced thrombocytopenia, current or any prior occurrences
* Known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or known hypersensitivity to heparin, aspirin, adenosine diphosphate (ADP) receptor inhibitors, or nitinol
* Known or suspected coagulopathy or abnormal coagulation parameters (defined as platelet count ≤ 100,000/mm³ or spontaneous International Normalized Ratio (INR) ≥1.5 in the absence of medication or known fibrinogen ≤1.5 g/L)
* Breastfeeding or pregnant
* Currently participating in active follow-up phase of another clinical study of an investigational drug or device
* Other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to provide written informed consent and/or to comply with study procedures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Safety | Perioperative/Periprocedural
  Rate of major device-related adverse events (MDRAEs), from device (Supira Introducer sheath) insertion through device removal (inclusive of Supira procedure-related serious adverse events [SAEs]).
Feasibility: | Perioperative/Periprocedural
  Successful hemodynamic support using the Supira System during high-risk percutaneous coronary intervention (HRPCI) and post-PCI as needed, with planned removal of the Supira Pump without the need to escalate/exchange to another MCS device such as Intra-aortic Balloon Pump (IABP) or Extracorporeal Membrane Oxygenation (ECMO).

SECONDARY OUTCOMES:
Secondary Study Endpoints | 30 days
  * Rate of technical success
  * Rate of procedural success
  * Rate of composite MDRAEs from cath lab discharge to Supira Catheter removal
  * Rate of composite MDRAEs from Supira Catheter removal to hospital discharge
  * Rate of MDRAEs from hospital discharge to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical, Study Director — Supira Medical
Locations (2):
- Georgia (2):
  - Tbilisi Heart and Vascular Clinic, Tbilisi, K'alak'i T'bilisi
  - Israeli-Georgian Medical Research Clinic HealthyCore 13g Tevdore-Mghvdeli Street Tbilisi Georgia, Tbilisi

IPD SHARING:
Plan to Share IPD: No